CLINICAL TRIAL: NCT02458794
Title: A Randomized Crossover Study of the LMA SupremeTM Versus Ambu-Aura GainTM in Adult Patients
Brief Title: Crossover Study of the LMA SupremeTM vs Ambu-Aura GainTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Schulthess Klinik (Other)
Collaborators: Krankenhaus Bozen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_5
Record Dates: First submitted 2015-05-20; First posted 2015-06-01 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Airway Morbidity
MeSH Terms: interventions — Platelet Function Tests

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA SupremeTM (Active Comparator): function tests: ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric tube insertion
  Interventions: Procedure: function tests; Device: LMA SupremeTM
- Ambu-Aura GainTM (Active Comparator): function tests: ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric tube insertion
  Interventions: Procedure: function tests; Device: Ambu-Aura GainTM

INTERVENTIONS:
Procedure: function tests — ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric tube insertion
Device: LMA SupremeTM
  Arms: LMA SupremeTM
Device: Ambu-Aura GainTM
  Arms: Ambu-Aura GainTM

SUMMARY:
The Ambu-Aura GainTM is a new extraglottic airway device which brings together features of both the LMA ProSealTM (high seal cuff, gastric access and bite block - to facilitate ventilation, airway protection and airway obstruction, respectively) and the LMA UniqueTM (single use - prevention of disease transmission). In the following randomized, crossover study, the investigators test the hypothesis that ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement differ between the Ambu-Aura GainTM and the LMA SupremeTM in paralyzed, anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Age 19-65 yr
* Written informed consent

Exclusion Criteria:

* Difficult airway
* Non fasted
* BMI > 35

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
oropharyngeal seal pressure | 5 minutes
  Oropharyngeal leak pressure was determined by closing the expiratory valve of the anesthesia breathing system and a fixed gas flow of 3 l minute-1. The airway pressure at which an equilibrium was reached was noted (maximum allowed 40 cm H2O).

SECONDARY OUTCOMES:
anatomic position | 5 minutes
  The anatomic position was assessed by passing a fiberoptic scope through the airway tube stopping 0,5 cm prior to the end of the tube. The airway tube view was scored using an established scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD MSc, Study Chair — Schulthess Klinik
Locations (2):
- Zentralkrankenhaus Bozen, Bolzano, Italy
- Schulthess Klinik, Zurich, Switzerland